CLINICAL TRIAL: NCT03088241
Title: Switch to Second-line Versus WHO-guided Standard of Care for Unsuppressed Patients on First-line ART With Viremia Below 1000 Copies/mL - a Multicenter, Parallel-group, Open-label, Randomized Clinical Study in Rural Lesotho
Brief Title: "Switch Either Near Suppression Or THOusand"
Acronym: SESOTHO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Niklaus Labhardt (Other)
Collaborators: Swiss Tropical & Public Health Institute (Other); SolidarMed, Lucerne, Switzerland (Unknown); SolidarMed (Other); University of Basel (Other); University Hospital, Basel, Switzerland (Other); Butha-Buthe Hospital, Lesotho (Unknown); Ministry of Health, Lesotho (Other Government)
Responsible Party: Sponsor-Investigator, Niklaus Labhardt, Niklaus Labhardt, MD MIH, Head of the research consortium, Swiss Tropical & Public Health Institute
Organization: Swiss Tropical & Public Health Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P002-17-1.0
Record Dates: First submitted 2017-03-12; First posted 2017-03-23 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: HIV/AIDS
Keywords: randomized clinical trial; low level viremia; lesotho; resource-limited setting; ART first-line failure
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: Multicenter (2-12 centers), parallel-group (1:1 allocation), open-label, superiority, prospective randomized clinical study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): switch to second-line ART
  Interventions: Other: switch
- Control (No Intervention): Standard of care: no switch to second-line ART

INTERVENTIONS:
Other: switch — switch to second-line ART
  Arms: Intervention

SUMMARY:
This trial addresses the question of the viral load (VL) threshold for switching from first-line to second-line antiretroviral therapy (ART). The WHO currently sets the threshold at 1000 copies/mL. However, the optimal threshold for defining virological failure and the need to switch ART regimen has not been determined. In fact, people with VL levels of less than 1000 copies/mL, however, not fully suppressed, are at increased risk for drug resistance mutations (DRM) and subsequent virological failure. In resource-limited settings where VL monitoring is not as frequent as in high-income countries, this could have serious implications and patients may continue on a failing regimen for a long period. Our research consortium will conduct a multicenter, parallel-group, open-label, randomized clinical trial in a resource-limited setting to assess whether a threshold of 100 copies/mL compared to the WHO-defined threshold of 1000 copies/mL for switching to second-line ART among unsuppressed HIV-positive patients on first-line ART will lead to better outcomes.

DETAILED DESCRIPTION:
Study background & rational:

The Joint United Nations Programme on HIV/AIDS (UNAIDS) launched the 90-90-90 targets for 2020 based on the result of newly-acquired scientific evidence that - irrespective of CD4 count - early antiretroviral treatment (ART) for HIV-positive individuals is beneficial to them and prevents HIV transmission. UNAIDS expects that the 90-90-90 targets will lead to a reduction in the yearly global HIV incidence from 2 million currently to 500,000 by 2020.

A crucial step to achieve the third pillar of the UNAIDS 90-90-90 targets - 90% viral suppression among HIV-positive individuals on treatment - and thus ensure a successful treatment outcome is the monitoring and management of first-line ART failure.

Since 2013, the WHO recommends routine viral load (rVL) measurement as the preferred monitoring strategy in resource-limited settings and defines virological failure as confirmed VL 1000 copies/mL despite good adherence. Specifically, the guidelines recommend that in case of a VL ≥ 1000 copies/mL the patient should undergo enhanced adherence support and a second VL test 3 months later. A second VL ≥ 1000 copies/mL with confirmed good adherence would trigger the switch to a second-line regimen, whereas if the VL is < 1000 copies/mL the patient should continue unaltered first-line ART. However, the optimal threshold for defining virological failure and the need for switching ART regimen has not yet been determined. In fact, people with VL levels of less than 1000 copies/mL, but not fully suppressed (usually defined as 50-100 copies/mL), are at a increased risk for drug resistance mutations (DRM) and subsequent virological failure. A recently published study from our research consortium in Lesotho indicates similar findings, demonstrating a significant accumulation of drug resistance mutations in patients with VL levels of less than 1000 copies/mL.

The VL threshold of 1000 copies/mL recommended by the WHO and the Lesotho national guidelines for the switch to second-line ART is likely to miss a substantial number of patients on first-line ART with persisting virus replication below 1000 copies/mL with DRM. In resource-limited settings where VL monitoring is not as frequent as in high-income countries, this could have serious implications: after a VL below 1000 copies/mL the patient may not receive a follow-up VL for up to a year, and thus may continue on a failing regimen for a long period of time. In conclusion, such patients are at increased risk for DRM, accumulation of further resistance mutations, drug-resistant virus transmission, and subsequent virological failure.

Study hypothesis:

Our research consortium hypothesizes that in patients on first-line ART with two consecutive unsuppressed VL measurements equal/more than 100 copies/mL, where the second VL is between 100 and 999 copies/mL, switch to second-line ART (intervention group) will lead to a higher rate of viral resuppression (VL < 50 copies/mL) and is therefore superior compared to not switching to second-line ART according to WHO guidelines (control group, standard of care).

Study design:

Multicenter (2-12 centers), parallel-group (1:1 allocation), open-label, superiority, prospective randomized clinical study.

ELIGIBILITY:
Inclusion Criteria:

* On NNRTI-based first-line ART with two consecutive unsuppressed VL equal/more 100 copies/mL, with the second VL between 100 and 999 copies/mL.
* Lives and/or works in the district of Butha-Buthe and declares to seek follow-up at one of the study-facilities
* Signed written informed consent. For children aged <16 years, a main caregiver, and for illiterate a literate witness, has to provide oral and written informed consent.

Exclusion Criteria:

* On ART less than 6 months
* On protease-inhibitor containing ART or any other second-line ART
* Bad adherence (self-reported at least 1 dose missing in the last 4 weeks, resp. 2 doses of a twice-daily-regimen)
* Clinical WHO stage 3 or 4 at enrolment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2020-05-23 (Actual); Study Completion 2020-05-23 (Actual)

PRIMARY OUTCOMES:
viral suppression | 9 months after randomization
  Proportion of virologically suppressed (VL < 50 copies/mL) participants 9 months after randomization.

SECONDARY OUTCOMES:
Proportion of participants with different VL thresholds (VL <100, <200, <400, <1000 copies/mL) at 9 months after randomization | 9 months after randomization
Adherence at 3, 6, 9 months, assessed by self-reported dose omission | 3, 6, 9 months after randomization
Change in values (versus values at baseline) of body-weight (kg) at 9 months | 9 months after randomization
Change in values (versus values at baseline) of haemoglobin (g/dL) at 9 months | 9 months after randomization
Change in values (versus values at baseline) of CD4 count (cells/mL) at 9 months | 9 months after randomization
Change in values (versus values at baseline) of lipids (total cholesterol, LDL, HDL, triglycerides; mmol/l) at 9 months | 9 months after randomization
Change in values (versus values at baseline) of new clinical WHO 3 or 4 events (proportion) count at 9 months | 9 months after randomization
Change in values (versus values at baseline) of deaths (all-causes) (proportion) at 9 months | 9 months after randomization
Proportion of patients with adverse events and serious adverse events at 9 months after randomization | 9 months after randomization
Long-term follow-up endpoint: Proportion of patients that are alive, retained in care and virologically suppressed (VL < 50 copies/mL) at 24 months | 24 months after randomization
Proportion of virologically suppressed (VL < 50 copies/mL) participants by demographic groups (children vs pregnant women vs adults) | 9 months after randomization
Proportion of virologically suppressed (VL < 50 copies/mL) participants by different VL groups at enrolment (VL 100-599 vs 600-999 copies/mL copies/mL) | 9 months after randomization
Proportion of participants with viral resuppression (<50 copies/mL) | 6 months after randomization
Sustained virologic failure | 6 and 9 months after randomization
  Proportion of participants with unsuppressed VL >50 copies/mL at 6 and 9 months

OTHER OUTCOMES:
Direct costs of each treatment arm | 9 months and 24 months after randomization
Prevalence of major viral resistance mutations to first-line regimen in each treatment arm for all samples for which an RT-PCR amplification is successful | 9 months after randomization
pre-specified subgroup: Log-drop | 9 months after randomization
  Viral resuppression among individuals with a >0.5 drop in log10 VL between the first screening VL and the second screening VL (i.e. VL at enrolment)

CONTACTS AND LOCATIONS:
Overall Officials: Niklaus Labhardt, MD MIH, Principal Investigator — Swiss Tropical and Public Health Institute, Basel
Locations (8):
- Lesotho (8):
  - Motebang Hospital, ART corner, Hlotse, Leribe District
  - Butha-Buthe Hospital, Butha-Buthe
  - Seboche Hospital, Butha-Buthe
  - Muela Health Center, Butha-Buthe
  - St. Paul Health Center, Butha-Buthe
  - St. Peters Health Center, Butha-Buthe
  - Senkatana ART clinic, Maseru
  - Mokhotlong Hospital, Mokhotlong

IPD SHARING:
Plan to Share IPD: Undecided
IPD (baseline characteristics, outcomes, follow-up data) will eventually be shared after completion of the study upon request.

REFERENCES:
- [Background] Amstutz A, Nsakala BL, Vanobberghen F, Muhairwe J, Glass TR, Achieng B, Sepeka M, Tlali K, Sao L, Thin K, Klimkait T, Battegay M, Labhardt ND. SESOTHO trial ("Switch Either near Suppression Or THOusand") - switch to second-line versus WHO-guided standard of care for unsuppressed patients on first-line ART with viremia below 1000 copies/mL: protocol of a multicenter, parallel-group, open-label, randomized clinical trial in Lesotho, Southern Africa. BMC Infect Dis. 2018 Feb 12;18(1):76. doi: 10.1186/s12879-018-2979-y. PMID 29433430
- [Result] Amstutz A, Nsakala BL, Vanobberghen F, Muhairwe J, Glass TR, Namane T, Mpholo T, Battegay M, Klimkait T, Labhardt ND. Switch to second-line versus continued first-line antiretroviral therapy for patients with low-level HIV-1 viremia: An open-label randomized controlled trial in Lesotho. PLoS Med. 2020 Sep 16;17(9):e1003325. doi: 10.1371/journal.pmed.1003325. eCollection 2020 Sep. PMID 32936795
- [Derived] Brown JA, Amstutz A, Nsakala BL, Seeburg U, Vanobberghen F, Muhairwe J, Klimkait T, Labhardt ND. Extensive drug resistance during low-level HIV viraemia while taking NNRTI-based ART supports lowering the viral load threshold for regimen switch in resource-limited settings: a pre-planned analysis from the SESOTHO trial. J Antimicrob Chemother. 2021 Apr 13;76(5):1294-1298. doi: 10.1093/jac/dkab025. PMID 33599270